CLINICAL TRIAL: NCT01963286
Title: Reduction of Inappropriate Shocks of Implantable Cardioverter Defibrillators (ICDs) With Enhanced SVT Discriminators
Acronym: ReduceIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-12-092-GE-HV
Record Dates: First submitted 2013-09-12; First posted 2013-10-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Tachycardia
Keywords: ICD; CRT-D; Sudden cardiac death; Device settings; Optimized programming strategy
MeSH Terms: conditions — Tachycardia; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enhanced SVT discriminators (Other): Patients with activated enhanced SVT discriminators (in accordance with predefined mandatory study settings)
  Interventions: Device: ICD with enhanced SVT discriminators

INTERVENTIONS:
Device: ICD with enhanced SVT discriminators — ICD will be programmed to uniform device settings with enhanced SVT discrimintators enabled.
  Other Names: Ellipse (St. Jude Medical); Fortify Assura (St. Jude Medical); Unify Assura (St. Jude Medical)

SUMMARY:
The purpose of this clinical investigation is the continued assessment of the decision accuracy of St. Jude Medical (SJM) ICD with enhanced SVT discriminators in the treatment of subjects with primary and secondary prevention of sudden cardiac death.

DETAILED DESCRIPTION:
With Ellipse™ and Fortify Assura™ ICD family, St. Jude Medical introduced enhanced device algorithms that may be helpful to further improve SVT discrimination success: SecureSense™, Far field morphology, Chamber Onset. These algorithms in combination with a tailored device setting (primary or secondary prevention) will be prospectively investigated within this trial.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or nonischemic cardiomyopathy
* Primary prevention or secondary prevention of Sudden cardiac death (SCD)
* Indication for ICD/CRT-D new implantation per current guidelines (1, 2, 3-chamber)
* The patient is ≥ 18 years of age
* The patient is able to understand the patient information and is capable to provide informed consent.
* The patient has provided written informed consent prior to any investigational related procedure

Exclusion Criteria:

* Previously implanted ICD/CRT-D
* Hypertrophic (with or without obstructive) cardiomyopathy
* Ion channel disorders (Long/Short-QT, Brugada syndrome etc…)
* New York Heart Association (NYHA) Class IV
* Recent cardiac decompensation (within previous 3 months)
* The patient is unable to comply with the follow up schedule.
* The patient is participating in another investigational device or drug investigation.
* The patient is pregnant or is planning to become pregnant during the duration of the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Inappropriate ICD shocks | 12 months
  Freedom from inappropriate automatically delivered ICD-shocks within 12 months Follow-Up (FU) period after ICD/CRT-D implantation

SECONDARY OUTCOMES:
ICD shocks for any reason | 12 months
  Freedom from automatically delivered ICD shocks for any reason during FU period
Inappropriate ICD therapies | 12 months
  Freedom from automatically delivered inappropriate ICD therapies during FU period
Untreated VT/VF | 12 months
  Freedom from untreated sustained ventricular tachycardia (VT) / ventricular fibrillation (VF) during FU period
Accuracy of ICD therapy decision | 12 months
  Accuracy of ICD therapy decision (VT/VF and nonVT/VF)
Specificity | 12 months
  Specificity for…
  * … other than sustained VT/VF
  * … SVT (Supraventricular tachycardia)
  * … different subtypes of SVTs (Sinus Tachycardia, Atrial Fibrillation, Atrial Flutter, other SVT).
Cardiac deaths | 12 months
  Cardiac deaths
Sensitivity | 12 months
  Sensitivity for sustained VT/VF
ICD/CRT-D related SAE | 12 months
  ICD/CRT-D related Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Johann C Geller, Prof. Dr., Study Chair — Zentralklinik Bad Berka
Locations (23):
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu
- Germany (21):
  - Praxis Dr. med. Bernhardt, Annaberg-Buchholz
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Hufeland Klinikum GmbH, Bad Langensalza
  - Caritas Krankenhaus, Bad Mergentheim
  - Medizinisches Versorgungszentrum am Küchwald GmbH, Chemnitz
  - Praxis Dr. med. Stellmach, Chemnitz
  - Klinikum Coburg GmbH, Coburg
  - Evangelisches Krankenhaus Kalk gGmbH, Cologne
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Oberhavel Kliniken GmbH Klinik Hennigsdorf, Hennigsdorf
  - Evangelisches Krankenhaus Holzminden gGmbH, Holzminden
  - Praxis Frau Dr. med. Gärtner, Leisnig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Klinikum Memmingen, Memmingen
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Christliches Krankenhaus Quakenbrück gGmbH, Quakenbrück
  - Gem.-Praxis Dres. med. Ebert / Stenzel, Riesa
  - Hegau-Bodensee-Klinikum mbH, Singen